CLINICAL TRIAL: NCT00018200
Title: Efficacy of Antidepressants in Chronic Back Pain
Brief Title: Effect of Antidepressants on Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADRD-018-98F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Back Pain; Sciatica
Keywords: analgesia; Back pain; sciatica
MeSH Terms: conditions — Back Pain; Sciatica; Agnosia | interventions — Desipramine; Clomipramine; Fluoxetine; Benztropine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): Desipramine, low, middle or high exposure
  Interventions: Drug: Desipramine
- Arm 2 (Experimental): Fluoxetine, low, middle, or high exposure
  Interventions: Drug: Fluoxetine
- Arm 3 (Placebo Comparator): Benztropine .125-.5mg daily
  Interventions: Drug: Benztropine

INTERVENTIONS:
Drug: Desipramine — Low exposure (40-70 ng/mL), Middle exposure (70-130 ng/mL), High exposure (130-200 ng/mL)
  Other Names: Anafranil
  Arms: Arm 1
Drug: Fluoxetine — Low exposure (200-399 ng/mL), Middle exposure (400-499 ng/mL), High exposure (500-700ng/mL)
  Other Names: Prozac
  Arms: Arm 2
Drug: Benztropine — Daily dose 0.125 to 0.5mg
  Other Names: Cogentin
  Arms: Arm 3

SUMMARY:
The purpose of this study is to determine whether different types of antidepressant medicines relieve back pain that has lasted at least six months on a daily basis. Study participants will be assigned to treatment with either a antidepressant acting on the serotonin system in the brain (fluoxetine), one acting on the noradrenaline system (desipramine, or to a control medication not expected to relieve pain (benztropine). Each participant will be seen at least nine times during their 12 weeks on medication. This is a phase 2/3, outpatient study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic back pain (pain on a daily basis for six months or longer)
* Age 18-65
* No major medical illness

Exclusion Criteria:

* medical contraindication to tricyclic antidepressants
* recent alcohol or substance use disorder
* bipolar disorder

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 1999-04; Primary Completion 2003-12 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Descriptor Differential Scale Pain Intensity | 12 weeks post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Joseph H. Atkinson, MD, Principal Investigator — VA San Diego Healthcare System, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, San Diego, California, United States

REFERENCES:
- [Result] Atkinson JH, Slater MA, Capparelli EV, Wallace MS, Zisook S, Abramson I, Matthews SC, Garfin SR. Efficacy of noradrenergic and serotonergic antidepressants in chronic back pain: a preliminary concentration-controlled trial. J Clin Psychopharmacol. 2007 Apr;27(2):135-42. doi: 10.1097/jcp.0b013e3180333ed5. PMID 17414235